CLINICAL TRIAL: NCT02360189
Title: Mechanisms of Social Inequalities in Post-hospitalization Rehabilitation in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Maria Pedersen, RN. MPH. Ph.D.-student, Nordsjaellands Hospital
Other Study IDs: ACS-12345
Record Dates: First submitted 2014-11-26; First posted 2015-02-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim: To identify psychological and socioeconomic predictors of cardiac-rehabilitation (CR) attendance and uncover mechanisms of CR non-attendance.

Design: Quantitative, observational, prospective study. Hypothesis a: Educational-level, comorbidity, anxiety, depression, self-efficacy, cohabitation and distance from residence are predictors of CR attendance.

Hypothesis b: The expected social gradient in CR attendance is explained partly by differential exposure of comorbidity, anxiety, depression, self-efficacy, cohabitation and distance to the rehabilitation clinic.

DETAILED DESCRIPTION:
Design: Quantitative, observational, prospective study. Self-administrated questionnaires, medical journals and telephone interviews will be used for data collecting.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with acute coronary syndrome (ACS) to Nordsjællands Hospital (ICD10: DI210-DI219, DI200, DI200B, DI200C, DI23, DI24) will be invited to participate in the survey as an ongoing process during the inclusion period (N=267).

Exclusion Criteria:

* Patients who are not able to submit written consent are excluded. Thus, patients with severe cognitive dysfunction or poor language skills are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized with acute coronary syndrome (ACS) to Nordsjællands Hospital (ICD10: DI210-DI219, DI200, DI200B, DI200C, DI23, DI24) will be invited to participate in the survey as an ongoing process during the inclusion period (N=267).
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2015-03; Primary Completion 2016-08 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Cardiac-rehabilitation attendance (yes/no) | 3 months post hospitalization

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Nordsjællands Hospital, Frederikssund., Frederikssund
  - Nordsjællands Hospital, Hillerød, Hillerød